CLINICAL TRIAL: NCT02235285
Title: Asian Outcomes of Primary Breast Augmentation in 162 Consecutive Cases Using Single Antibiotic Breast Irrigation by A Single Surgeon Under Sedative Anesthesia (Propofol Infusion)
Brief Title: Asian Outcomes of Primary Breast Augmentation
Acronym: BA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Winners Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Breast Augmentarion
Record Dates: First submitted 2014-09-05; First posted 2014-09-09 (Estimated); Results first posted 2015-09-21 (Estimated); Last update posted 2018-05-04 (Actual); Status verified 2018-05

CONDITIONS: Breast Augmentation
Keywords: capsular contracture; reoperation; breast augmentation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- breast augmentation,reoperation (Experimental): A retrospective chart review was performed to examine a total of 162 patients received the same brand of implants for primary breast augmentation under sedative anesthesia (propofol infusion) in a single surgeon's practice.
  Interventions: Procedure: primary breast augmentation

INTERVENTIONS:
Procedure: primary breast augmentation — With the patient under sedative anesthesia, wide preparation and draping by using povidone-iodine are performed with using talc-free gloves and povidone-iodine gauze nipple shields. Tumescent solution is infiltrated in the precise plane. Pockets are developed precisely with blunt dissection with fingers and instruments under both direct and indirect visions simultaneously, if needed, with using endoscopy, while careful hemostasis done. After dissection, two pockets are irrigated with 300ml of single antibiotic solution without active evacuation of the irrigation. When re-draping and re-preparation by using povidone-iodine are performed before implant insertion, a new pair of talc-free gloves is used and cleansed with the single antibiotic solution.

SUMMARY:
In 162 Asian patients, primary breast augmentations were performed by a single surgeon during 5 years. The purpose of this study evaluates Asian outcomes in primary breast augmentation using single antibiotic breast irrigation by a single surgeon's practice and examines the comparison of Asian and Western outcomes in primary breast augmentation.

DETAILED DESCRIPTION:
A retrospective chart review was performed to examine a total of 162 patients received the same brand of implants for primary breast augmentation under sedative anesthesia (propofol infusion) in a single surgeon's practice. Asian patients' demographics, preoperative and postoperative measurements, surgical technique (single antibiotic breast irrigation), implant type, size, texture, soft tissue coverage, implant placement, incision approach, complications, and incidence of reoperation were documented.

ELIGIBILITY:
Inclusion Criteria:

* primary case

Exclusion Criteria:

* secondary case
* breast reduction

Ages: 22 Years to 57 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 162 (Actual)
Dates: Start 2010-01; Primary Completion 2014-04 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: CHEOLHWAN KIM, M.D., Principal Investigator — Winners Clinic
Locations (1):
- The Department of Plastic Surgery, Winners Clinic, Seoul, South Korea

REFERENCES:
- [Background] Spear SL, Murphy DK, Slicton A, Walker PS; Inamed Silicone Breast Implant U.S. Study Group. Inamed silicone breast implant core study results at 6 years. Plast Reconstr Surg. 2007 Dec;120(7 Suppl 1):8S-16S. doi: 10.1097/01.prs.0000286580.93214.df. PMID 18090808

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Retrospective analysis was performed on 162 patients undergoing primary breast augmentation by a single surgeon during a 5-year period from 2010 to 2015.
Pre-assignment Details: This study presents data for 162 primary breast augmentation in either alone (n=152; 93.82 percent) or in conjunction with mastopexy (n=9; 5.56 percent) and inverted nipple correction (n=1; 0.62 percent) .
Groups:
- Breast Augmentation,Reoperation: The most common cause of reoperation in breast augmentation is a capsular contracture. So the prevention of capsular contracture is very important in breast augmentation. The investigators reviewed 162-consecutive patients underwent breast augmentation by one surgeon. The rate of follow-up at 5 years for all patients was 92 percent.
Period: Overall Study
Arm/Group | Breast Augmentation,Reoperation
Started | 162
Completed | 149
Not Completed | 13

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Participants were 162-consecutive patients underwent primary breast augmentation by one surgeon.
Arm/Group | All Study Participants
Number analyzed (Participants) | 162
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 162
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.98 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 162
  Male | 0
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 162

OUTCOME MEASURES:

1. Primary Outcome: Post Surgical Complications and Reoperation Rate During Breast Augmentation
Description: The investigators reviewed 162-consecutive patients underwent breast augmentation by one surgeon for reoperation rate.
Time Frame: 5 years
Measure: Mean (Standard Deviation); unit: percentage of participants
Groups:
- Breast Augmentation, Reoperation: The investigators reviewed 162-consecutive patients underwent breast augmentation by one surgeon for reoperation rate.
Arm/Group | Breast Augmentation, Reoperation
Number analyzed (Participants) | 162
percentage of participants
  reoperation rate | 1.85 (0.05)
  complications | 1.85 (0.05)

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Breast Augmentation, Reoperation
Serious Adverse Events (participants affected / at risk) | 3/162
Other Adverse Events (participants affected / at risk) | 0/162
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Breast Augmentation, Reoperation (N=162)
Capsular contracture (Skin and subcutaneous tissue disorders) | 2
Rippling (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes